CLINICAL TRIAL: NCT04468074
Title: Study on the Use of Virtual Reality Neuropsychological Therapy Technology (VRNT) for Chronic Back Pain
Brief Title: Virtual Reality Treatment for Adults With Chronic Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CognifiSense Inc. (Industry)
Collaborators: University of Colorado, Boulder (Other); National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 19-0526; 1R43NR017575-01A1 (NIH)
Record Dates: First submitted 2020-06-30; First posted 2020-07-13 (Actual); Results first posted 2022-06-23 (Actual); Last update posted 2022-06-23 (Actual); Status verified 2022-05

CONDITIONS: Chronic Pain; Back Pain Lower Back Chronic; Back Pain
MeSH Terms: conditions — Chronic Pain; Back Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Therapy Group (Experimental): Therapy Group participants start the treatment period with three 1 ½ hour introductory sessions:
  1. An education session on the science behind chronic pain and a basic overview of the VR therapy.
  2. A session to customize the VR experience to match the participant's own pain experience.
  3. A training session on the use of the VR hardware and software.
  Upon completion, participants begin using the VR therapy app at home once a day, 5 times a week (minimum), for a total of 8 weeks. The VR app contains different training exercises. A workbook provides a schedule and background on each of the training sessions.
  Therapy Group participants may continue their other pain treatment regimes, and are asked to notify the research team of any changes.
  Interventions: Device: Virtual Reality Therapy for Chronic Pain
- Standard of Care (SOC) Group (No Intervention): The SOC Group (no-intervention) completes a daily pain survey. SOC Group participants are asked to maintain their pain treatment regimes, and are asked to notify the research team of any changes.

INTERVENTIONS:
Device: Virtual Reality Therapy for Chronic Pain — 1. A 1 1/2 PowerPoint-based education session on the science behind chronic pain and a basic overview of the VR therapy
  2. Virtual Reality Therapy: a virtual reality therapy consisting of different psychological training exercises
  Other Names: Virtual Reality Neuropsychological Therapy (VRNT)
  Arms: Therapy Group

SUMMARY:
Participants with chronic back pain will complete an online eligibility questionnaire. After signing a consent form, eligible participants enter a two-week baseline period ("Baseline Period") during which they complete a daily pain survey. Following the Baseline Period all participants complete an MRI scan. After the MRI, scan participants are randomized into a treatment group ("Therapy Group") or a no-intervention group ("Standard of Care Group" or "SOC Group") with a ratio of 1:1 (treatment:SOC). Therapy Group participants receive education about chronic pain. They also participate in sessions to personalize their Virtual Reality (VR) experience, and to complete training on the use of the VR hardware and software. Therapy Group participants complete the treatment for 8 weeks ("Therapy Period"), after which they return the VR equipment. All participants take a second MRI scan approximately 8-weeks after the first MRI; for the Therapy Group this is at the end of the Therapy Period. After the Therapy Period, Therapy Group participants continue to complete daily pain surveys during a two-week follow-up period ("Follow-Up Period"). All participants complete self-reported clinical outcomes and behavioral measures surveys before and after the Baseline Period, 4 weeks after the first MRI (for Therapy Group this is mid-way through the Therapy Period), and before and after the Follow-Up Period. For Therapy Group participants the study ends with the final surveys and an exit interview at the end of the Follow-up Period. Study Extension (Add-on): SOC Group participants may receive the treatment after the Follow-Up period. Those who elect to do so will complete the same set of surveys as the Therapy Group did during the treatment phase; however, since there is no comparison group, data from this study extension is not used in the main outcomes analyses.

ELIGIBILITY:
Inclusion Criteria:

* Participants aged 21 to 70 with Chronic Back Pain.
* Chronic Back Pain will be defined according to criteria established by recent NIH task force. Pain duration must be ≥ 3 months, with back pain being an ongoing problem for at least half the days of last 6 months; i.e., either pain every day for past 3 months, or half or more of the days for past 6+ months.
* Subjects must rate pain intensity at ≥ 4/10 on Brief Pain Inventory (average pain over the last week).
* Participants must also be comfortable and able to communicate via email, text message, or phone in English. Participants must also be comfortable using a video-conferencing service such as Zoom to complete the on-line sessions.

Exclusion Criteria:

* Applicants, who are pregnant, planning pregnancy, or breastfeeding
* Back pain associated with compensation / litigation within 1 year.
* Leg pain greater than back pain (suggests neuropathic pain; may be less responsive to psychological therapy).
* Chronic pain other than chronic back pain.
* Diagnoses of schizophrenia, multiple personality dissociative identity disorder.
* History of major depressive disorder not controlled with medication or other conditions that produce significant cognitive or emotional disability.
* History of substance abuse.
* Inability to undergo MRI (determined at screening; see XVI: Risks to Participants).
* Any clinically significant unstable medical abnormality or acute or chronic disease of cardiovascular, gastrointestinal, respiratory (e.g., chronic obstructive pulmonary disease), hepatic, or renal systems; including: history of cardiovascular disease or issues (e.g., recent heart attack), stroke; brain surgery, or brain tumor; Diabetes; cancer (last 12 months); diagnosis of a specific inflammatory disorder: rheumatoid arthritis, polymyalgia rheumatica, scleroderma, Lupus; polymyositis; or Cauda Equina syndrome.
* History of seizure disorder, epilepsy, convulsions, or increased intracranial pressure anytime except pediatric febrile seizures.
* History of vertigo, dizziness, susceptibility to motion sickness
* History of head injury within 6 months,
* Unexplained, unintended weight loss of 'â• 20 lbs in past year.
* Self-reported history of (digital) eye strain or computer vision syndrome.
* Unable or unwilling to meet study attendance requirements.
* MRI contraindications as determined by MRI safety screen (e.g., pregnancy, metal in body, claustrophobia, using the standard screen conducted by the MRI imaging facility).

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2020-06-09 (Actual); Primary Completion 2021-04-13 (Actual); Study Completion 2021-06-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marta Ceko, Ph.D., Principal Investigator — University of Colorado, Boulder; Lynn Webster, MD, Principal Investigator — CognifiSense Inc.; Tassilo Baeuerle, Principal Investigator — CognifiSense Inc.
Locations (1):
- University of Colorado, Boulder, Boulder, Colorado, United States

REFERENCES:
- [Background] Cherkin DC, Sherman KJ, Balderson BH, Cook AJ, Anderson ML, Hawkes RJ, Hansen KE, Turner JA. Effect of Mindfulness-Based Stress Reduction vs Cognitive Behavioral Therapy or Usual Care on Back Pain and Functional Limitations in Adults With Chronic Low Back Pain: A Randomized Clinical Trial. JAMA. 2016 Mar 22-29;315(12):1240-9. doi: 10.1001/jama.2016.2323. PMID 27002445
- [Derived] Ceko M, Baeuerle T, Webster L, Wager TD, Lumley MA. The effects of virtual reality neuroscience-based therapy on clinical and neuroimaging outcomes in patients with chronic back pain: a randomized clinical trial. Pain. 2024 Aug 1;165(8):1860-1874. doi: 10.1097/j.pain.0000000000003198. Epub 2024 Mar 8. PMID 38466872

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited via online (e.g., social media) advertising between December 2019 and September 2020. The first participant was enrolled on June 9, 2020, and the last participant was enrolled in October 2020.
Pre-assignment Details: Of 1,346 applicants, 270 met inclusion criteria. Of these, 72 were enrolled in the study; however, 11 withdrew before start / randomization. 61 participants started the study (completed randomization). After a 2-week baseline period, participants were randomized into the Experimental and No Intervention Groups.
Groups:
- Therapy Group: Therapy Group participants start the treatment period with three 1 ½ hour introductory sessions:
  1. An education session on the science behind chronic pain and a basic overview of the VR therapy.
  2. A session to customize the VR experience to match the participant's own pain experience.
  3. A training session on the use of the VR hardware and software.
  Upon completion, participants begin using the VR therapy app at home once a day, 5 times a week (minimum), for a total of 8 weeks. The VR app contains different training exercises. A workbook provides a schedule and background on each of the training sessions.
  Therapy Group participants may continue their other pain treatment regimes, and are asked to notify the research team of any changes.
  Virtual Reality Therapy for Chronic Pain: 1) A 1 1/2 PowerPoint-based education session on the science behind chronic pain and a basic overview of the VR therapy 2) Virtual Reality Therapy: a virtual reality therapy consisting of different psychological training exercises
Period: Overall Study
Arm/Group | Therapy Group | Standard of Care (SOC) Group
Started | 31 | 30
Completed | 30 | 30
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Therapy Group | Standard of Care (SOC) Group | Total
Number analyzed (Participants) | 31 | 30 | 61
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.1 (10) | 33.5 (9.2) | 34.2 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 15 | 30
  Male | 16 | 15 | 31
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 2 | 5
  Not Hispanic or Latino | 24 | 23 | 47
  Unknown or Not Reported | 4 | 5 | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 2
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 1 | 2 | 3
  White | 28 | 26 | 54
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Change in Pain Intensity and Interference.
Description: Brief Pain Inventory-short form (BPI-SF). Measured on Scale of 0 to 10, 0 = no pain, 10 = worst pain imaginable.
Time Frame: Change from pre-treatment to post-treatment = 8 weeks.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Therapy Group | Standard of Care (SOC) Group
Number analyzed (Participants) | 30 | 30
units on a scale | -1.5 (1.7) | -0.5 (1.3)
Statistical Analysis 1: Comparison: Therapy Group vs Standard of Care (SOC) Group; Test type: Superiority; p = 0.014, Mixed Models Analysis; Mean Difference (Net) = 1

2. Secondary Outcome: Change in Quality of Life.
Description: Quality of Life (HRQoL SF-12) Questionnaire: yes / no questions and 3-point / 6-point Likert Scale questions; e.g., 1 = [negative impact] all of the time (worse outcome), 6 = [negative impact] none of the time. HRQoL results in two sub-scales / components (Physical and Mental). The mean of these was taken to result in a single value.
Time Frame: Baseline (average of survey data at beginning and end of a 2-week baseline period) and at the end of the 8 week therapy / control period.
Population: Intent to Treat
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Therapy Group | Standard of Care (SOC) Group
Number analyzed (Participants) | 30 | 30
units on a scale | 3.68 (4.7) | .89 (3.5)
Statistical Analysis 1: Comparison: Therapy Group vs Standard of Care (SOC) Group; Test type: Superiority; p = 0.0159, Mixed Models Analysis; Mean Difference (Net) = 2.79

3. Secondary Outcome: Change in Back Pain Disability.
Description: Oswestry Low Back Pain Disability Questionnaire (OLBPD). 6-point Likert Scale questions on impact of pain on various life aspects; e.g., 1 = no negative impact, 6 = prevents normal activity (worse outcome). Participants completed questionnaire at the beginning and end of a 2-week baseline period and at the end of the 8 week therapy / control period. The starting values were the average of the two reported pain measures at the beginning and end of the baseline period
Time Frame: Change from pre-treatment to post-treatment = 8 weeks.
Population: Intent to treat
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Therapy Group | Standard of Care (SOC) Group
Number analyzed (Participants) | 30 | 30
units on a scale | -4.22 (6.2) | -.37 (4.5)
Statistical Analysis 1: Comparison: Therapy Group vs Standard of Care (SOC) Group; Test type: Superiority; p = 0.0066, Mixed Models Analysis; Median Difference (Net) = -3.85

4. Other Pre Specified Outcome: Change in Pain Bothersomeness.
Description: Pain Bothersomeness Scale. 0-10 scale: 0 = not at all bothersome; 10 = extremely bothersome) (Source: Cherkin et al. 2016).
Time Frame: Change from pre-treatment to post-treatment = 8 weeks.
Reporting Status: Not Posted

5. Other Pre Specified Outcome: Change in Medications and Therapies.
Description: A questionnaire asking participants to list the type and dosage / frequency of medication and therapies the participant is using for their back pain and for any other medical conditions. The list and dosage of medications and the type and frequencies of therapies will be compared pre- and post-treatment (8-week interval) to assess change in other pain therapies.
Time Frame: Change from pre-treatment to post-treatment = 8 weeks.
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Change in Pain Catastrophizing.
Description: Pain Catastrophizing Questionnaire (PCS). 4-point Likert scale: = not at all, 4 = all the time (worse outcome).
Time Frame: Change from pre-treatment to post-treatment = 8 weeks.
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Change in Fear of Pain.
Description: Fear of Pain Questionnaire. 5-point Likert scale: = not at all, 5 = extreme (worse outcome).
Time Frame: Change from pre-treatment to post-treatment = 8 weeks.
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Change in Fear of Movement.
Description: Tampa Scale of Kinesiophobia (TSK). 4-point Likert scale: = strongly disagree, 4 = strongly agree (worse outcome).
Time Frame: Change from pre-treatment to post-treatment = 8 weeks.
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Change in Sleep Quality.
Description: Patient Reported Outcomes Measurement Information System (PROMIS) short form for Sleep Disturbance: 8 items. 5-point Likert scales: 5 = not at all, 1 = very much (worse outcome).
Time Frame: Change from pre-treatment to post-treatment = 8 weeks.
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Change in Fatigue Symptoms.
Description: Patient Reported Outcomes Measurement Information System (PROMIS) short form for Fatigue: 8 items. 5-point Likert scales: 1 = not at all, 5 = very much (worse outcome).
Time Frame: Change from pre-treatment to post-treatment = 8 weeks.
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Change in Depression.
Description: Patient Reported Outcomes Measurement Information System (PROMIS) short form for Depression: 8 items. 5-point Likert scales: 5 = never, 1 = always (worse outcome).
Time Frame: Change from pre-treatment to post-treatment = 8 weeks.
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Change in Pain Attitudes.
Description: Survey of Pain Attitudes (SOPA) Short Form. 6-point Likert scale: 5 = This is very untrue for me, 1 = This is very true for me [worse outcome].
Time Frame: Change from pre-treatment to post-treatment = 8 weeks.
Reporting Status: Not Posted

13. Other Pre Specified Outcome: Change in Self-efficacy.
Description: General Self-Efficacy Scale. 4-point Likert scale: 1 = not at all true [worse outcome], 4 = exactly true.
Time Frame: Change from pre-treatment to post-treatment = 8 weeks.
Reporting Status: Not Posted

14. Other Pre Specified Outcome: Expectations of Treatment Success.
Description: Expectations of Treatment Success Survey. 0 to 10 scale: 0 = none, 10 = most (best outcome).
Time Frame: Before Therapy Period begins (pre-treatment; after 2-week baseline).
Reporting Status: Not Posted

15. Other Pre Specified Outcome: Impression of Treatment Success.
Description: Patient Global Impression of Change (PGIC). 7-point scale: 0 = no change (condition has got worse [worst outcome]), 10 = a great deal better, and a considerable improvement that has made all the difference.
Time Frame: At the end of the Therapy Period (post-treatment; approx. 10 weeks into study).
Reporting Status: Not Posted

16. Other Pre Specified Outcome: Change in Optimism
Description: Life Orientation Test (LOT-R). 5-point Likert scale: 0 = strongly disagree, 4 = strongly agree (worse outcome is a function of the question).
Time Frame: Change from pre-treatment to post-treatment = 8 weeks.
Reporting Status: Not Posted

17. Other Pre Specified Outcome: Change in Emotion Regulation.
Description: Emotion Regulation Questionnaire (ERQ). 7-point Likert scale: 1 = strongly disagree, 7 = strongly agree (worse outcome is a function of the question).
Time Frame: Change from pre-treatment to post-treatment = 8 weeks.
Reporting Status: Not Posted

18. Other Pre Specified Outcome: Change in Mindfulness.
Description: Mindful Attention Awareness Scale (MAAS). 7-point Likert scale: 0 = almost always (worse outcome), 7 = almost never.
Time Frame: Change from pre-treatment to post-treatment = 8 weeks.
Reporting Status: Not Posted

19. Other Pre Specified Outcome: Change in Pain Coping Strategies.
Description: Coping Strategies Questionnaire (CSQ). 7-point Likert scale: 0 = never do, 7 = always do that (worse outcome is a function of the question).
Time Frame: Change from pre-treatment to post-treatment = 8 weeks.
Reporting Status: Not Posted

20. Other Pre Specified Outcome: Change in Structural (Brain) MRI.
Description: Acquire 2 structural MRI brain scans (before and after treatment) to measure brain gray matter changes due to treatment.
Time Frame: Change from pre-treatment to post-treatment = 8 weeks.
Reporting Status: Not Posted

21. Other Pre Specified Outcome: Change in Resting-State Functional MRI.
Description: Acquire 2 functional MRI brain scans (before and after treatment), during which the participants will rest, to measure functional brain changes due to treatment.
Time Frame: from pre-treatment to post-treatment = 8 weeks.
Reporting Status: Not Posted

22. Other Pre Specified Outcome: Change in Diffusion Tensor Imaging (DTI) MRI.
Description: Acquire 2 DTI MRI scans (before and after treatment) to measure brain white matter changes due to treatment.
Time Frame: Change from pre-treatment to post-treatment = 8 weeks.
Reporting Status: Not Posted

23. Other Pre Specified Outcome: Assessment of Usability of VR Device.
Description: Questionnaire with 10 questions on usability of the VR device; 5-point Likert scale: 1 = strongly disagree, 5 = strongly agree (worse outcome is a function of the question).
Time Frame: At the end of the Therapy Period (post-treatment; approx. 10 weeks into study).
Reporting Status: Not Posted

24. Other Pre Specified Outcome: Assessment of Sense of Presence in the VR Environment.
Description: Questionnaire with 14 questions about the participant's sense of presence in the virtual environment - based on IGP Presence Questionnaire; 5-point Likert scale: 1 = fully disagree, 5 = fully agree (worse outcome is a function of the question).
Time Frame: At the end of the Therapy Period (post-treatment; approx. 10 weeks into study).
Reporting Status: Not Posted

25. Other Pre Specified Outcome: Assessment of Sense of Embodiment in the VR Environment.
Description: Questionnaire with 10 questions about the participant's sense of embodiment in the virtual reality environment - based on the Gonzalez-Franko Embodiment Questionnaire; 7-point Likert scale from -3 = strongly disagree to +3 = strongly agree (worse outcome is a function of the question).
Time Frame: At the end of the Therapy Period (post-treatment; approx. 10 weeks into study)
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 8 weeks
Arm/Group | Therapy Group | Standard of Care (SOC) Group
All-Cause Mortality (participants affected / at risk) | 0/31 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/30
Other Adverse Events (participants affected / at risk) | 0/31 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2020-08-29): https://cdn.clinicaltrials.gov/large-docs/74/NCT04468074/Prot_003.pdf
  • Statistical Analysis Plan (2022-04-12): https://cdn.clinicaltrials.gov/large-docs/74/NCT04468074/SAP_004.pdf
  • Informed Consent Form (2020-06-19): https://cdn.clinicaltrials.gov/large-docs/74/NCT04468074/ICF_000.pdf